CLINICAL TRIAL: NCT05970133
Title: Functional Recovery and Oncologic Efficacy of Robotic Versus Laparoscopy NOSE for Patients With Stage I III Left Sided Colon Cancer: A Randomized Controlled Trial
Brief Title: Robotic Versus Laparoscopy NOSE for Stage I-III Left-sided Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301224RINB
Record Dates: First submitted 2023-07-18; First posted 2023-08-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Natural orifice specimen extraction; Laparoscopic surgery; Robotic surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic surgery (Experimental): The patients in this group will undergo laparoscopic surgery.
  Interventions: Procedure: Colectomy with NOSE procedure
- Robotic surgery (Active Comparator): The patients in this group will undergo robotic surgery.
  Interventions: Procedure: Colectomy with NOSE procedure

INTERVENTIONS:
Procedure: Colectomy with NOSE procedure — The specimen will be extract from the anus.

SUMMARY:
In this project, the investigator aims to provide the level 1 evidence for the comparison of robotic versus laparoscopic NOSE for the surgery of stage I-III colorectal cancer. the investigator hypothesize that, with the increased maneuverability of the current robotic system, robotic surgery will be a good option for patients with stage I-III colorectal cancer requiring a NOSE procedure.

DETAILED DESCRIPTION:
Over the past three decades, laparoscopic surgery has evolved incessantly, especially in the field of colorectal surgery. It has been widely accepted by surgeons and patients in light of the better peri-operative outcomes and analogical long-term effectiveness, compared with open surgery for colorectal cancers. However, current conventional laparoscopic colorectal surgery requires an additional abdominal incision for specimen retrieval and sometimes for intestinal reconstruction, which increases the risk of various postoperative complications, including pain, surgical site infection, incisional hernia, and injury to the epigastric artery and abdominal cutaneous nerves, and, consequently, can delay postoperative chemotherapy.

To mitigate these unfavorable outcomes, natural orifice specimen extraction (NOSE) via the anus, stomach, or vagina, was introduced. One randomized trial reported better short-term surgical outcomes, including reduced pain and lower analgesia requirements for laparoscopic NOSE colectomy, compared with conventional laparoscopic colectomy. Transanal specimen extraction has been utilized after laparoscopic colon or rectal cancer surgery and has been found to be feasible, safe, and oncologically sound in selected cases. Several multiport laparoscopic platforms are currently available to complete all NOSE procedures and reestablish intestinal continuity with a single stapled anastomosis, which has been shown to improve short-term results compared with conventional laparoscopic colectomy. However, concerns remain regarding the long-term oncologic safety (tumor cell spillage with local recurrence and long-term survival) when NOSE is used for colorectal malignancy.

A barrier to wider adoption of NOSE is technical difficulty. The mini-laparotomy, in some cases, is used to perform a majority of the operation, as in hand-assisted laparoscopy. Adoption of NOSE by surgeons who typically perform colectomies in this fashion would be faced with a steeper learning curve than surgeons who use the mini-laparotomy solely as a specimen extraction site. On that note, intracorporeal anastomosis is a prerequisite skill for those adopting NOSE. Removal of more proximal specimens, as in a right colectomy, requires the presence of a skilled endoscopist who can snare and pull the specimen endoluminally through the length of the distal gastrointestinal tract. Specimen extraction via the vagina requires a posterior colpotomy, an operative maneuver that is not typically performed by general or colorectal surgeons. Furthermore, these technical challenges are amplified by a lack of standardization of the technique.

The demands for these technical skills are more important in removing right-sided colon pathology, as compared to left-sided pathology. There are inherent anatomic factors that make NOSE for right-sided colon pathology more difficult. Right colectomy specimens extracted through the lower gastrointestinal tract via distal colotomy must travel the length of the remaining transverse, descending, and sigmoid colon, through the rectum and out of the anus using an endoscope. While this was demonstrated to be feasible in 2010 by Eshuis et al, it is inherently difficult due to the anatomically narrow and torturous sigmoid colon. In that series, extraction via colotomy failed in 2 of 10 patients due to the bulk of the specimen. This technique is still performed in some centers, though limitations related to the size of the specimen are stricter than for left-sided colon lesions. This approach has little practicality due to its significant technical challenges, hence its limited use.

Bacterial contamination is always a concern during the NOSE procedure. Most researchers strongly suggest that mechanical bowel preparation, intraoperative transanal lavage with povidone iodine solution, transluminal wound protector, and prophylactic antibiotics are applied to reduce the bacterial load. Recently, a study showed that the risk of bacterial contamination with NOSE was not significantly higher than that in conventional laparoscopic surgery. In some studies, patients who had NOSE did not experience significant postoperative morbidity or laboratory data changes, such as leukocytosis, CRP level elevation, rectal wound-related complications or leakage, than the conventional group.

Tumor size is considered before applying the NOSE procedure. Many authors limit indications to tumors smaller than 3 - 6.5 cm. Some authors have stated that obese patients are not suitable for transrectal specimen extraction and set the BMI cutoff at > 28-35 kg/m2. Most researchers considered patients with a bulky mesocolon, a narrow pelvis, and previous pelvic surgery with severe adhesions were not eligible for NOSE.

It is generally accepted that laparoscopic NOSE can achieve oncological and surgical safety comparable to that of conventional laparoscopic surgery for patients with sigmoid and rectal cancer. Remarkably, Laparoscopic NOSE patients were associated with a shorter hospital stay, shorter time to first flatus or defecation, less postoperative pain, and fewer surgical site infections and total perioperative complications. In general, the operative time in laparoscopic NOSE was longer than that in conventional laparoscopic surgery. The long-term oncological efficacy of laparoscopic NOSE seems to be equivalent to that of conventional laparoscopic surgery. Furthermore, specimen retrieval through alternative routes to avoid an abdominal incision is beneficial for the prevention of incisional hernia.

Currently, robotic surgical approaches are becoming more popular for treating colorectal cancer. Robotic techniques can overcome some technical limitations of laparoscopic surgery, including an unstable camera view and straight laparoscopic instruments. Robotic surgery is advantageous because it provides surgeon-control of the camera, high-definition three-dimensional vision, excellent ergonomics, decreased physiological tremor, more freedom of angles of instruments, and the ability to simultaneously control the camera and two additional instruments that facilitate traction and countertraction, all of which enable to facilitate the procedures, even in difficult settings.

The unique advantages of the surgical robot make colorectal surgery operations more precise and intelligent, providing more options for minimizing operative stress during colorectal surgery. The proximity between the sigmoid colon and rectum to the anal location provides a favorable predisposition for transanal specimen retrieval without significantly increasing the difficulty of the surgical operation. However, to date, only very few studies compared robotic NOSE versus laparoscopic NOSE for the surgery of colorectal cancer. Actually, our preliminary data has shown the safety and feasibility of robotic NOSE, as compared with laparoscopic NOSE for the surgery of colorectal cancer.

Even to date, laparoscopic NOSE procedure for colorectal cancer is still not popular due to the technique difficulty associated with an intra-corporeal anastomosis for NOSE and the oncologic concern of tumor spillage at the staple line during tumor retrieval process. In this respect, the introduction of robotic system can overcome the technical difficulties.

In this project, the investigator aims to provide the level 1 evidence for the comparison of robotic versus laparoscopic NOSE for the surgery of stage I-III colorectal cancer. the investigator hypothesize that, with the increased maneuverability of the current robotic system, robotic surgery will be a good option for patients with stage I-III colorectal cancer requiring a NOSE procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Primary colon cancers located at the left sided colonic anatomic location, including distal transverse colon, colonic splenic flexure, descending colon, sigm oid descending colonic junction, sigmoid colon and upper rectum that required the mobilization of colonic splenic flexure to facilitate a curative resection and trans anal specimen extraction ;
2. TNM Stage I III adenocarcinomas;
3. Curative and elective surgery;
4. American Society of Anesthesiology (ASA) class I to III patients;
5. Age >18 years.

Exclusion Criteria:

1. Cecal, ascending, the proximal and middle transverse colon cancers; and the middle or lower rectal cancers;
2. Emergency or palliative surgery;
3. Evidence of disseminated disease or adjacent organ invasion;
4. Primary tumor mass >8 cm in diameter;
5. Morbidly obese patients, that is, body mass index (BMI) ≥40 kg/m 2 ;
6. Previous major surgery of upper abdomen or pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
The surgical efficiency of both NOSE procedures | Intraoperative hours with an average of 5 hours
  The operation time defined as the incision of wound and application of the surgical dressing

SECONDARY OUTCOMES:
Overall disease-free survival | 5 years
  The duration between surgery and death
Overall recurrence-free survival | 5 years
  The duration between surgery and recurrence
Incontinence | 6 months
  Evaluated by questionnaire
Time to return work | 1 year
  Disability
Total fee and equipment fee | 3 months
  Total Cost
Blood loss | Intraoperative hours with an average of 5 years
  measured by the amount Mof blood in suction bottle and the number of blood soaked gauzes
Conversion rate | Intraoperative hours with an average of 5 years
  Conversion from robotic surgery to laparoscopic surgery or open surgery
Complications | 30 days
  Any complication during or after surgery grading by Calvien -Dindo classification
Wound size | Intraoperative hours with an average of 5 years
  Total length of the wounds
Serum C reactive protein (CRP) | Throughout the admission with an average of 7 days
  CRP could be an indicator of the severity of surgical stress.
Erythrocyte sedimentation rate (ESR) | Throughout the admission with an average of 7 days
  ESR could be an indicator of the severity of surgical stress.
Blood lymphocyte counts | Throughout the admission with an average of 7 days
  Blood lymphocyte counts could be an indicator of the severity of surgical stress.
CD4+ to CD8+ ratio | ESR could be an indicator of the severity of surgical stress.
  CD4 to CD8 ratio could be an indicator of the severity of surgical stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan